CLINICAL TRIAL: NCT03524378
Title: Chronic Low Back Pain in Seafood Workers: a Pilot Intervention Study to Identify Modifiable Work and Movement Solutions
Brief Title: Modifiable Work and Movement Solutions Low Back Pain in Seafood Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201702245 - N; 3U54OH011230-02S1 (NIH); 6U54OH011230-05M002 (NIH)
Record Dates: First submitted 2018-04-20; First posted 2018-05-14 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Chronic Low Back Pain
Keywords: repetitive strain; ergonomics; participatory ergonomics; chronic low back pain; seafood workers
MeSH Terms: interventions — Ergonomics

STUDY DESIGN:
Intervention Model Description: Within-subject control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ergonomic and movement modifications (Other): No group assignment - all participants will self select suitable ergonomic or movement modifications
  Interventions: Behavioral: Ergonomic and movement modifications

INTERVENTIONS:
Behavioral: Ergonomic and movement modifications — Introduction of basic ergonomic and self-management principles, participants will review video clips of the prioritized and revised solutions. Adjustments in work tasks, movement strategies or self-management techniques will be self selected by workers after an educational session using videotapes of work processes.

SUMMARY:
Chronic low back pain has been identified as a major problem for seafood and agricultural workers, and is known to affect worker health and productivity. The aims of this study are to: 1) identify modifiable, sector-specific, work and movement solutions with the potential to reduce the burden or severity of chronic lower back pain in clam workers and 2) determine the extent that participants adopt identified solution(s), and the impact on functional difficulty and low back pain.

DETAILED DESCRIPTION:
This pilot/feasibility pre-post intervention study will use a participatory ergonomic approach without a control group or randomization. The participatory approach will foster capacity building by creating support within the workplace communities and by involving seafood workers in developing context specific solutions for their own work practice, increasing the potential for adoption and success.

Phase 1: Specific Aim 1: Identify modifiable, sector-specific work and movement solutions with that can reduce the burden or severity of chronic lower back pain

1. Development of rapid prototype video clips: clam workers will be videotaped performing typical work tasks during daily operations on the boat, as well as transporting, sorting and packing clams will be analyzed. Key movements and positions such as lifting, prolonged static flexed positions that may be contributing to repetitive stress in the low back region will be categorized. Short clips will be edited to create examples of movements and positions for each category potentially contributing to low back pain.
2. Prioritization of specific tasks and relevant solutions by key leaders: Up to 10 participants with a history of chronic low back pain for more than 3 months will be recruited by the Cedar Key Aquaculture Association for the initial pilot testing of research methods. Once participants have provided informed consent, they will complete a general demographic survey, functional disability and pain questionnaire and surveys to measure co-variates that include pain fear and anxiety, self-efficacy and coping questions.

Focus groups will be held in the participant's work settings with consented individuals from the same work teams to ensure application within a specific context and promote discussion directed towards the best outcomes. Participants will discuss major tasks and factors contributing to their low back pain using the video clips to target discussions and their opinions of options that would help alleviate or prevent pain. Only clips from the relevant teams will be used for each focus group. The focus groups will be recorded and transcribed for analysis and as a record of discussion.

Basic principles of ergonomic adaptation and movement modification for repetitive work activities on and off the boat and lifting will be introduced using demonstrations and discussion in a small group format. Participants will discuss other possible solutions. Self-management including movement strategies and pain relief techniques will be introduced and demonstrated by the principal investigator. The educational session will be videotaped to ensure all relevant discussions are considered during the development of interventions and to assist with reliability of intervention delivery.

At the end of the focus group and educational session, participants will prioritize their most problematic work tasks and most relevant and feasible solutions. In a follow up visit, participants will be videotaped demonstrating the tasks and selected methods to reduce or prevent repetitive stress determined from the focus group. With permission from the participants, selected videos will be edited to provide clips to be used in subsequent workshops. Only participants who agree to be videotaped for educational purposes will be included in this session.

Phase II: Specific Aim 2: Determine the extent that participants adopt identified solution(s), and the impact of their self-selected work and movement modifications on their functional difficulty in the workplace related to low back pain.

In addition to the workers recruited for specific aim 1, up to 24 additional clam workers for a total of up to 34 participants will be recruited with the same criteria; chronic low back pain for more than 3 months, over the age of 18 and employed full time in clam gathering/preparation.

1. Baseline: Once participants have provided informed consent, they will complete a general demographic survey, functional disability and pain questionnaire and surveys to measure co-variates that include pain fear and anxiety, self-efficacy and coping questions. Functional disability, pain reports and work related functional ability will be recorded once a week for 4 weeks.
2. Implementation of interventions, focus group discussion and identification of individual solutions: After the baseline period, workers will contribute to small focus groups of 4-6 individuals in their work team. After introduction of basic ergonomic and self-management principles, participants will review video clips of the prioritized and revised solutions identified in Specific Aim 1. After indicating their preferences, the feasibility of solutions will be discussed. Following this discussion, participants will indicate if they believe that the adjustments in work tasks, movement strategies or self-management apply to their work, are easy to implement and are likely to decrease their back pain. Workers will suggest any additional options to implement the ergonomic principles. At the end of the focus group, participants will select 3 options to use in their work activities for 8 weeks.
3. Follow up: The research team will contact participants by text or phone once a week to provide reminders. At 4 weeks the initial survey data will be repeated. The frequency and consistency of use of the solutions during work activities will be reported to reflect adoption, along with any pre-post changes in measures. After completion of the 8 weeks, individuals will also comment on the effectiveness, feasibility and impact of solutions on their low back pain and job performance. Participants will also be asked to suggest options for implementation and provide feedback on how to optimize the intervention for wider dissemination, and if they would recommend the solutions to co-workers.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic low back pain
* Employed full time in clam harvesting/processing

Exclusion Criteria:

* History of spinal surgery in past 3 years
* Recent hospitalization in the past year for any condition
* Subjects currently seeking disability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Patient Specific Functional Scale | Change from baseline average measured over 4 weeks, after 4 and 8 weeks
  3 work items regarded as the most painful or difficult activities will selected by each participant and rated on a 0-100 scale with inability to complete a task rated as 0/100 and ability to perform the activity without any difficulty due to low back pain as a 100/100. Participants will also report the amount of time that they are able to complete the task without stopping or changing tasks due to low back pain for each activity.
Pain rating scales | Change from baseline average measured over 4 weeks, after 4 and 8 weeks
  Pain ratings for each of the items identified in the patient specific functional scale (best, worst and average ratings) over the past day with 0/100 reflecting no pain, 100/100 most excruciating pain possible

SECONDARY OUTCOMES:
Short form pain anxiety symptom scale | Baseline, Day 1, 4 weeks, 8 weeks
  Self reported survey to reflect anxiety (Ranges from 0-5 with 5 being always in pain)
Fear avoidance single item question | Baseline, Day 1, 4 weeks, 8 weeks
  Single item question to reflect fear avoidance measured as both a co-variate or possible outcome
Pain self-efficacy questions | Baseline, Day 1, 4 weeks, 8 weeks
  Two questions to reflect fear avoidance measured as both a co-variate or outcome
Pain coping questions | Baseline, Day 1, 4 weeks, 8 weeks
  Two questions to reflect fear avoidance measured as both a co-variate or outcome
Oswestry Disability Index for low back pain | Baseline, at 4 weeks and after intervention at 8 weeks
  Modified Oswestry Disability Index is a valid and reliable self reported instrument reflecting disability related to low back pain. Ten items related to difficulty with activities of daily living are scored on a 0-5 scale, 0 representing no difficulty, 5 representing the greatest disability. An index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. 0-20% is considered minimal disability; 21%-40%: moderate disability:41%-60%: severe disability: 61%-80%: extremely severe disability; 81%-100%:complete disability

OTHER OUTCOMES:
Adoption of strategies | 8 weeks
  Number of individuals adopting work-related methods for more than 50% of the time

CONTACTS AND LOCATIONS:
Overall Officials: Kim Dunleavy, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Cedar Key Aquaculture Association, Cedar Key, Florida
  - UF Health, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dunleavy K, Kane A, Coffman A, Reidy J, Bishop MD. Outcomes of Participatory Ergonomics and Self-management in Commercial Clam Farmers with Chronic Low Back Pain: A Feasibility Study. J Agromedicine. 2022 Apr;27(2):217-231. doi: 10.1080/1059924X.2021.2004961. Epub 2021 Nov 23. PMID 34772318